CLINICAL TRIAL: NCT06523244
Title: Comparison of Photo Disinfection With Chitosan Nanoparticles Enriched ICG Over ICG as an Adjunct to Open Flap Debridement in Stage II/III Grade B/C Periodontitis. RCT
Brief Title: Comparing Photodisinfection of Chitosan NP Enriched ICG Over ICG as Adjunct to OFD: RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02_D012_00046
Record Dates: First submitted 2024-07-19; First posted 2024-07-26 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Periodontal Pocket
MeSH Terms: conditions — Periodontal Pocket | interventions — Photochemotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test group (Experimental): PDT with chitosan nanoparticles enriched ICG
  Interventions: Procedure: PHOTODYNAMIC THERAPY
- Control group (Active Comparator): PDT with ICG
  Interventions: Procedure: PHOTODYNAMIC THERAPY

INTERVENTIONS:
Procedure: PHOTODYNAMIC THERAPY — Respective photosensitive dye solution is applied on to the surgical site, including all the root surfaces. Vacuum suction is used to remove the excess dye from the site and to prevent ingestion of the dye solution The dye is activated with 810nm diode laser with continuous wave frequency and power of 0.3 W with 400 µm fiber tip for 20 seconds/spot. After this, the area is irrigated with saline.

SUMMARY:
The current study is a prospective randomised study-Comparison of photodisinfection with chitosan nanoparticles enriched indocyanine green over indocyanine green as an adjunct to open flap debridement in the management of stage II/III grade B/C periodontitis.

DETAILED DESCRIPTION:
A total of 24 patients fulfilling inclusion criteria will be randomly assigned into two treatment groups (Test and Control). Open flap debridement followed by photodynamic therapy using dyes is carried out.

Test group (n=12) - PDT with Chitosan nanoparticles enriched ICG Control group(n=12) - PDT with ICG Microbial levels of P.gingivalis is analysed with PCR analysis on baseline and 3 months after intervention.

ELIGIBILITY:
Inclusion criteria:

* Systemically healthy subjects
* Age group 30-55yrs.
* Diagnosed with Stages II/III grade B/C periodontitis.
* Presenting with persistent pocket depth ≥5mm after initial non-surgical therapy.
* Optimal plaque control
* Good compliance

Exclusion criteria:

* Subjects on antibiotic therapy within last six months of enrollment
* Previous history of periodontal surgery
* Allergy to drugs and materials used in this study
* Pregnant woman
* Subjects with deleterious habits like smoking, tobacco chewing.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
MICROBIAL ANALYSIS | 3 MONTHS
  LEVELS OF P. GINGIVALIS